CLINICAL TRIAL: NCT00120016
Title: Design and Feasibility of a Mediterranean Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 051517; 03B043-REV
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: cancer prevention; diet; nutrition; polyunsaturated fat; olive oil
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mediterranean diet
  Interventions: Behavioral: dietary counseling
- 2 (No Intervention): non-intervention diet

INTERVENTIONS:
Behavioral: dietary counseling — telephone counseling
  Other Names: high MUFA diet
  Arms: 1

SUMMARY:
Epidemiological observations indicate that a Greek-Mediterranean dietary pattern has great potential for cancer prevention, but more definitive data on the preventive effects of this diet are needed. Two distinct aspects of this eating pattern are the type of fat consumed and a high fruit/vegetable intake. If the diet is feasible, it could be used in future clinical trials of breast cancer prevention. In this study, women randomly receive either a control diet or an intervention diet for 6 months. The intervention diet replaces half of the typical American fat intake with foods such as olive oil and nuts. The fruit and vegetable goal is 7-9 servings/day and includes several categories of fruits, vegetables, and herbs. Blood samples are drawn and analyzed for fatty acids derived from fats, micronutrients from fruits and vegetables, and markers of oxidative stress. This dietary trial will provide important data on the ability of women following typical American eating patterns to change their dietary intakes to reflect a Greek-Mediterranean pattern.

DETAILED DESCRIPTION:
It has been difficult to identify specific nutrients or food groups associated with breast cancer risk from epidemiological studies done in the U.S. Attention is now turning to the importance of overall eating patterns. A Greek-Mediterranean dietary pattern has great potential for cancer prevention. Two distinct aspects of this eating pattern are the type of fat consumed and a high fruit/vegetable intake relative to average intakes in the United States. We propose to develop and test an exchange list Greek-Mediterranean diet that could be used in future clinical trials of breast cancer prevention in women at increased risk. In this proposed study, women will be randomized to either continue their own usual diet or follow an intervention diet for 6 months. The intervention diet will be designed to decrease polyunsaturated (P) and saturated (S) fat intakes while increasing monounsaturated (M) fat intake. The P:S:M ratio of a typical American diet is about 1.0:1.5:1.7, and the goal for this intervention diet will be 1:2:5, which is much closer to that of the traditional Greek diet. A predominant source of fat will be olive oil. The fruit and vegetable goal will be 7-9 servings/day, depending on energy intake. These dietary changes will be achieved using individualized telephone counseling and a monthly group session with a dietitian. Menus will be provided as examples, but the diets will be self-selected. Compliance to the dietary goals will be assessed by food records and levels of plasma fatty acids, lipids and carotenoids. As a feasibility investigation for the planning of larger trials, plasma 8-isoprostane, oxidized lycopene, insulin and glucose levels will also be assessed since these may lend insight into two possible mechanisms that may be responsible for the cancer preventive effects of this diet. This dietary trial will provide important data on the ability of women following typical American eating patterns to change their dietary intakes to reflect a Greek-Mediterranean pattern. This intervention approach can then be tested for its effects on markers of breast cancer risk in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Normal weight
* Age 25-65
* Monounsaturated fat intake less than 48% of total fat
* Fruit and vegetable intake less than 5.5 servings/day
* Total fat intake more than 23% of energy

Exclusion Criteria:

* High blood pressure
* Obese
* Pregnant or lactating
* On medically prescribed diets
* Taking supplements that obscure the effects of diet
* Diabetes

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
fatty acid intakes | 6 months
carotenoids intakes | 6 months
fatty acid ratios in blood | 6 months
carotenoids in blood | 6 months
cholesterol in blood | 6 months

SECONDARY OUTCOMES:
markers of oxidative stress in blood | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Djuric Z, Ren J, Blythe J, VanLoon G, Sen A. A Mediterranean dietary intervention in healthy American women changes plasma carotenoids and fatty acids in distinct clusters. Nutr Res. 2009 Mar;29(3):156-63. doi: 10.1016/j.nutres.2009.03.001. PMID 19358929
- [Result] Djuric Z, Vanloon G, Radakovich K, Dilaura NM, Heilbrun LK, Sen A. Design of a Mediterranean exchange list diet implemented by telephone counseling. J Am Diet Assoc. 2008 Dec;108(12):2059-65. doi: 10.1016/j.jada.2008.09.006. PMID 19027409